CLINICAL TRIAL: NCT06550674
Title: Identification of New Candidate Genes for Hereditary Predisposition to Uveal Melanoma
Acronym: IGCMU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: Association Nationale des Patients atteints de cancers de l'oeil (A.N.P.A.C.O.) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A00030-47
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma; hereditary predisposition; candidate genes identification
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- constitutional genetic analysis (Experimental): Constitutional genetic exome analysis will be performed on the blood sample. If necessary, an analysis on a second independent sample (jugal smear) will be carried out if a probably pathogenic or pathogenic variant in a hereditary cancer predisposition gene is identified.
  Interventions: Genetic: Constitutional exome analysis

INTERVENTIONS:
Genetic: Constitutional exome analysis — For each patient included:
  * A family tree is drawn up, reporting personal and family histories of cancer. The patient's anatomopathological reports, related to his or her tumor lesions, are retrieved, in order to confirm/clarify individual or family diagnoses.
  * A blood sample and a jugal smear are taken to enable constitutional genetic exome analysis for research purposes.

SUMMARY:
Only 20% of familial uveal melanomas are explained by a hereditary predisposition, implying the presence of as yet unknown hereditary predispositions. This hypothesis is reinforced by epidemiological studies revealing an excess risk of prostate cancer, thyroid cancer and leukemia in patients who have developed uveal melanoma, even though these cancers are not part of the tumor spectrum of known hereditary predispositions to uveal melanoma (BAP1, MBD4). The identification of new candidate genes, once validated, would enable us to offer these families appropriate surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a personal history of uveal melanoma (newly diagnosed, under treatment or in follow-up)
* Enrolled in or benefiting from a social security scheme

Exclusion Criteria:

* Causal pathogenic variation identified in BAP1 or MBD4
* Patient does not consent to constitutional genetic analysis for diagnostic purposes
* Patient not consenting to a constitutional genetic analysis for research purposes
* Pregnant and breast-feeding women
* Patients under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Identify new candidate genes for hereditary cancer predisposition in patients with uveal melanoma by constitutional exome analysis | At baseline
  Variants of interest are selected from the data using the following filter:
  * Variant with frequency < 1% (GnomAD)
  * Shared by at least 2 sufferers in the cohort
  * Truncating (nonsense, with frame shift, on a canonical splice site -2, -1 and +1 +2)
  * Missense from a list of "cancer" genes and Combined Annotation Dependent Depletion (CADD) score > 20 (COSMIC Tier1 and Tier2)
  Variants will be interpreted using various databases and prediction tools:
  * Functions: genecards, pubmed, uniprot
  * Expression profiles: cbioportal, GEPIA
  * For splice variants: CADD, Splice AI
  * For exonic variants: CADD, SIFT, Polyphene

SECONDARY OUTCOMES:
Explore genes known to be involved in other cancer predisposition already described in the occurrence of uveal melanoma, but whose association has not yet been established with certainty. | At baseline
  Number of patients with a mutation on BRCA1, BRCA2, CHEK2, PALB2, POT1, MSH6 or MLH1

CONTACTS AND LOCATIONS:
Overall Officials: Mathis LEPAGE, Dr, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean PERRIN, Clermont-Ferrand, Puy-de-Dôme, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Godiveau M, Ginzac A, Bidet Y, Ponelle-Chachuat F, Privat M, Durando X, Cavaille M, Lepage M. Identification of new candidate genes for the hereditary predisposition to uveal melanoma: IGCMU trial. Front Oncol. 2025 Jan 24;15:1538924. doi: 10.3389/fonc.2025.1538924. eCollection 2025. PMID 39926282